CLINICAL TRIAL: NCT03237351
Title: Goal Directed Fluid Therapy Guided Fluid Management in Pneumoresection: a Randomized Controlled Trial
Brief Title: Goal Directed Fluid Therapy Guided Fluid Management in Pneumoresection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZhiHeng Liu (Other)
Responsible Party: Sponsor-Investigator, ZhiHeng Liu, Chair of Department of Anesthesiology, Shenzhen Second People's Hospital
Organization: Shenzhen Second People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017041102
Record Dates: First submitted 2017-07-24; First posted 2017-08-02 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Goal-directed Fluid Therapy
Keywords: goal-directed fluid therapy; thoracic surgery, video-assisted; acute lung injury
MeSH Terms: conditions — Acute Lung Injury | interventions — Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional therapy group (Active Comparator): Patients in Conventional therapy group were received fluid therapy: intraoperative transfusion volume=maintenance fluids+deficit replacement+restoration of losses and with heart rate, mean arterial pressure, urine measurement ect.
  Interventions: Device: Fluid therapy
- Low value of PPV group (Experimental): Patients in low value of PPV group were received fluid therapy according to PPV (3% ≤PPV < 5%) .
  Interventions: Device: Fluid therapy
- High value of PPV group (Experimental): Patients in high value of PPV group were received fluid therapy according to PPV (5% ≤PPV < 8%) .
  Interventions: Device: Fluid therapy

INTERVENTIONS:
Device: Fluid therapy — Conventional therapy group: conventional arterial blood pressure monitoring. Low value of PPV group and high value of PPV group:pulse pressure variation monitoring with arterial blood pressure monitoring.

SUMMARY:
Perioperative fluid management is a key component of anesthetic management during thoracic surgery. On one hand, fluid restriction could compromise perfusion of vital organs and surgical anastomosis. On the other hand, fluid overload could lead to cardiopulmonary complications, notably pulmonary edema, which carries a high mortality rate. Perioperative fluid management to avoid postpneumonectomy pulmonary edema has been previously reviewed. Therefore, to achieve the balance between preventing fluid overload and optimising organ perfusion, the practical index to guide fluid management, which can predict whether fluid loading will improve haemodynamic conditions in an individual patient, would be very valuable during lung surgery. Perioperative goal-directed fluid therapy (GDFT) is a cornerstone of tissue perfusion and oxygenation, and it can improve surgical outcomes. Respiratory variations of arterial pressure [i.e. pulse pressure variation (PPV) and systolic pressure variation] can predict fluid responsiveness in mechanically ventilated patients under various conditions. Therefore, pressure variations are increasingly being advocated for fluid management.This study will discuss the effects of pulse pressure variation(PPV) in different level during anesthesia on patients with oxygenation index and short-term prognosis undergoing video-assisted thoracoscopic surgery for pneumoresection.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I-III; aged 18-60 years old; BMI 18.5 ~ 28 kg/m2

Exclusion Criteria:

* Refused to participate in the experiment, hepatic/renal/cardiac dysfunction, severe valvular disease, frequent arrhythmia, moderate anemia and severe electrolyte disturbance before operation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Oxygenation Index in 48 hours | Before induction, 5 minutes before the end of one-lung ventilation, 48 hours after the operation

SECONDARY OUTCOMES:
The duration of surgery | During surgery period
The duration of mechanical ventilation | During surgery period
Crystalloid administered | During surgery period
Colloid administered | During surgery period
Blood loss | During surgery period
Urine output | During surgery period
Number of patients received vasopressor | During surgery period
Blood pressure | Before the surgery and 48 hours after surgery
Leukocyte | Before the surgery and 48 hours after surgery
Hematocrit | Before the surgery and 48 hours after surgery
Complication until hospital discharge | 1 month after surgery
Hospital stay postoperatively | 1 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giglio MT, Marucci M, Testini M, Brienza N. Goal-directed haemodynamic therapy and gastrointestinal complications in major surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2009 Nov;103(5):637-46. doi: 10.1093/bja/aep279. PMID 19837807
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Background] Ripolles-Melchor J, Espinosa A, Martinez-Hurtado E, Abad-Gurumeta A, Casans-Frances R, Fernandez-Perez C, Lopez-Timoneda F, Calvo-Vecino JM. Perioperative goal-directed hemodynamic therapy in noncardiac surgery: a systematic review and meta-analysis. J Clin Anesth. 2016 Feb;28:105-15. doi: 10.1016/j.jclinane.2015.08.004. Epub 2015 Oct 2. PMID 26440438
- [Background] Chau EH, Slinger P. Perioperative fluid management for pulmonary resection surgery and esophagectomy. Semin Cardiothorac Vasc Anesth. 2014 Mar;18(1):36-44. doi: 10.1177/1089253213491014. Epub 2013 May 29. PMID 23719773
- [Background] Zhang J, Chen CQ, Lei XZ, Feng ZY, Zhu SM. Goal-directed fluid optimization based on stroke volume variation and cardiac index during one-lung ventilation in patients undergoing thoracoscopy lobectomy operations: a pilot study. Clinics (Sao Paulo). 2013 Jul;68(7):1065-70. doi: 10.6061/clinics/2013(07)27. PMID 23917675
- [Background] Lee JH, Jeon Y, Bahk JH, Gil NS, Hong DM, Kim JH, Kim HJ. Pulse pressure variation as a predictor of fluid responsiveness during one-lung ventilation for lung surgery using thoracotomy: randomised controlled study. Eur J Anaesthesiol. 2011 Jan;28(1):39-44. doi: 10.1097/EJA.0b013e32834089cf. PMID 21088596